CLINICAL TRIAL: NCT05807035
Title: A Phase I Trial of Autologous Tumour Vaccine for Advanced Solid Cancers
Brief Title: Autologous Tumour Vaccine Trial
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Vaxine Pty Ltd (Industry)
Collaborators: Australian Respiratory and Sleep Medicine Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CAN001
Record Dates: First submitted 2023-03-28; First posted 2023-04-10 (Actual); Last update posted 2025-09-17 (Actual); Status verified 2025-09

CONDITIONS: Solid Tumor
Keywords: cancer; tumor; immunotherapy; vaccine; neoplasm
MeSH Terms: conditions — Neoplasms | interventions — FANG vaccine

STUDY DESIGN:
Intervention Model Description: All subjects ewill receive active intervention in an n=1 study design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Radvax (Experimental): This is a single arm study where all participants will get active Radvax autologous tumour vaccine weekly for 4 weeks and then monthly thereafter
  Interventions: Biological: Radvax

INTERVENTIONS:
Biological: Radvax — Vaccine extracted from patient's own tumour tissue formulated with polysaccharide adjuvant
  Other Names: Autologous tumor vaccine

SUMMARY:
Phase 1 trial to evaluate the feasibility of preparation, safety, tolerability and response to a personalised autologous tumour vaccine (ATV) formulated with Advax adjuvant when administered to patients with advanced solid cancers either as monotherapy or in combination with other standard of care agents

DETAILED DESCRIPTION:
Radvax is a newly developed vaccine where extracted autologous tumour proteins are combined with the non-inflammatory Advax delta inulin adjuvant. Cancer immunotherapy has had a renewed interest due to the recent success and regulatory approval of immune checkpoint inhibitors and CAR-T cells. However, only a proportion of cancer patients derive benefit from these agents and hence there is an ongoing need to improve outcomes of patients with advanced solid tumours. Radvax is a novel simplified ATV approach whereby soluble tumour antigens are extracted from tumour samples obtained at surgery or from biopsy and formulated with Advax adjuvant. This vaccine has shown efficacy in murine models of glioma and pancreatic cancer, clinical trials of canine cancer patients. Radvax is now being assessed in a Phase 1 clinical trial of advanced solid cancers. Autologous tumour vaccines (ATV) will be generated from surgically removed or biopsied fresh tumour tissue. ATV is manufactured as a tumour lysate extract which is stored frozen, and then formulated with Advax adjuvant on day of administration. Doses of ATV will be administered on days 1, 8, 15, 22 during cycle 1 and then 4 weeks thereafter until total of up to 12 cycles Primary Endpoint(s): Incidence of grade 3 or 4 adverse effects Secondary Endpoint(s): Response rates by iRECIST, progression free survival and overall survival Exploratory Endpoints: To study parameters and predictive biomarkers of cancer response

ELIGIBILITY:
Inclusion Criteria:

* Subjects must have histologically or cytologically confirmed advanced solid cancers or hematological cancers (lymphomas only)
* Subjects must have received at least one prior therapy for this disease, with the exception that subjects for whom no standard therapy options exist or who decline standard therapies can be considered for inclusion after discussions with the investigator team.
* Performance status ≤ 2 (ECOG performance status)
* Subjects or their parents if a child must have the ability to understand and the willingness to sign a written informed consent document.
* If no suitable cancer tissue is already available to make the vaccine, to be enrolled in the trial participants must be willing to undergo surgery and/or fresh tumour biopsy to obtain tissue to allow the preparation of the vaccine and their primary care team needs to have agreed to perform these procedures for them to obtain tumour tissue. The trial team will provide advice on appropriate tissue collection and arrange transport and processing but are not responsible for arranging such surgery or paying for its cost.

Exclusion Criteria:

* Subjects receiving any other investigational agents within the preceding 4 weeks.
* Pregnant women because of the unknown risk of adverse events in the foetus secondary to treatment of the mother with ATV.
* Any potential participant where suitable cancer tissue is not available for preparation of the vaccine
* Any condition that the Investigator deems may make a potential participant unsuitable for entry into the trial.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-02-10 (Actual); Primary Completion 2026-02-10 (Estimated); Study Completion 2028-02-10 (Estimated)

PRIMARY OUTCOMES:
Incidence of grade 3 or 4 adverse effects | Interval from time of vaccination to 7 days post vaccination
  Incidence of grade 3 or 4 adverse effects related to vaccine administration

SECONDARY OUTCOMES:
Progression free survival | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 60 months
  Progression free survival
Overall survival | From date of randomization to date of death from any cause, assessed up to 60 months
  Overall survival
Response rate by RECIST version 1.1 | From date of randomization, assessed each 6 months up to 60 months
  modified Response Evaluation Criteria in Solid Tumours (RECIST version 1.1) in cancer immunotherapy trials

CONTACTS AND LOCATIONS:
Overall Officials: Dimitar Sajkov, MBBS/PhD, Principal Investigator — ARASMI
Locations (1):
- ARASMI, Adelaide, South Australia, Australia

IPD SHARING:
Plan to Share IPD: No